CLINICAL TRIAL: NCT01806584
Title: A Phase 2, Single-blind, Randomized, Controlled, Multi-center Study to Evaluate the Efficacy and Safety of SRM003 (Vascugel®) in the Treatment of Subjects With Vascular Injury Resulting From Arteriovenous Graft Surgery for Hemodialysis Access
Brief Title: An Efficacy and Safety Study of SRM003 in the Treatment of Subjects Undergoing Placement of an Arteriovenous Graft to Facilitate Hemodialysis Access
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Development of SRM003 was discontinued based on portfolio prioritization.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AVG01-SRM003
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Results first posted 2015-12-31 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Arteriovenous Graft
Keywords: Vascular Injury; Arteriovenous Graft Surgery; Hemodialysis Access
MeSH Terms: conditions — Vascular System Injuries | interventions — Gelatin Sponge, Absorbable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SRM003 (Active Comparator)
  Interventions: Biological: SRM003
- Participating Site's standard practice (Other)
  Interventions: Other: Participating Site's standard practice

INTERVENTIONS:
Biological: SRM003 — One time implant (3 SRM003 pieces) on surgery day.
  Other Names: Allogeneic human aortic endothelial cells cultured in a gelatin matrix (Gelfoam®).
  Arms: SRM003
Other: Participating Site's standard practice — Subjects will receive sites' standard practice treatment during the surgical procedure
  Arms: Participating Site's standard practice

SUMMARY:
A study to evaluate the efficacy of SRM003 treatment versus participating sites' standard practice treatment in extending the duration of primary patency after arteriovenous graft surgery in subjects with end-stage renal disease.

It is hypothesized that when placed outside the blood vessel, the seeded SRM003 gelatin matrix containing endothelial cells can provide a continuous supply of multiple growth regulatory compounds to the underlying cells within the blood vessel, while being protected from the effects of blood flow in the vessel(s) or complications resulting from being in direct contact with the point of injury.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18 years of age or older at the time of signing and dating informed consent (no upper age limit), can be male or female.
2. Subject who is of child bearing potential must agree to use adequate contraception for 6 months after randomization.
3. Subject must be currently undergoing hemodialysis or anticipating the start of hemodialysis and must require a new permanent prosthetic expanded polytetrafluoroethylene AVG placed in the upper extremity.
4. Subject must have a life expectancy of at least 78 weeks after randomization.
5. Subject must be able to understand and be willing to complete all study requirements.

Exclusion Criteria:

1. Subject is currently on an active organ transplant list from a deceased donor or is undergoing assessment and expects to be placed on the active organ or bone marrow transplant list within the next 78 weeks from surgery, or expects to receive a living donor organ or bone marrow within the next 78 weeks and is unwilling to change transplant list status to "hold" for 3 months after randomization.
2. Subject has had more than 3 access placement surgeries (defined as a new access, not a revision) in the target limb.
3. Subject has medical conditions and diseases that may cause non-compliance with the protocol
4. Subject has a known allergy to bovine/porcine products or collagen/gelatin products.
5. Subject has a history of intravenous drug use within 6 months prior to screening
6. Subject is morbidly obese, defined as having a body mass index >40.
7. Pregnant or nursing woman, or plans to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-03-28 (Actual); Primary Completion 2014-10-23 (Actual); Study Completion 2014-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (46):
- United States (46):
  - Akdhc Medical Research Services, Phoenix, Arizona
  - Tucson Vascular Consultants, Tucson, Arizona
  - Ladenheim Dialysis Access Center, Fresno, California
  - California Institute of Renal Research, La Mesa, California
  - VA Long Beach Health Care System Pharmacy, Long Beach, California
  - The Regents University of California Los Angeles, Los Angeles, California
  - California Institute of Renal Research, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Tampa General Hospital, Tampa, Florida
  - Georgia Regents University, Augusta, Georgia
  - Illinois Kidney Disease & Hypertension Center, Peoria, Illinois
  - University of Louisville, Louisville, Kentucky
  - Ochsner Baptist Medical Center, Clinical Trials Unit, New Orleans, Louisiana
  - Louisiana State University Health Science Center Shreveport, Shreveport, Louisiana
  - Baystate Medical Center Pharmacy, Springfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Renaissance Renal Research Institute, LLC, Detroit, Michigan
  - McLaren Northern Michigan Hospital-NISUS Research, Petoskey, Michigan
  - Providence Hospital, Research Dept., Southfield, Michigan
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Sierra Nevada Nephrology Consultants, Reno, Nevada
  - United Health Services, Johnson City, New York
  - Mount Sinai School of Medicine Lab, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Metrolina Nephrology Associates, PA, Charlotte, North Carolina
  - ECU Department of Nephrology and Hypertension, Greenville, North Carolina
  - Sanford Research/USD-Fargo, Fargo, North Dakota
  - University of Cincinnati Physicians Company, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Kaiser Permanente Northwest, Milwaukie, Oregon
  - Northwest Renal Clinic, Inc., Portland, Oregon
  - Penn Medicine, Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Delaware Valley Nephrology and Hypertension Associates, PC, Philadelphia, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - SC Nephrology & Hypertension Center, Inc., Orangeburg, South Carolina
  - Erlanger Hospital Pharmacy, Chattanooga, Tennessee
  - Nephrology Associates, P.C., Nashville, Tennessee
  - Baylor College of Medicine ICTR, Houston, Texas
  - Fletcher Allen Health Care Renal Service, Burlington, Vermont
  - Sentara Vascular Specialists, Norfolk, Virginia
  - University of Wisconsin, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Participating Site's Standard Practice: Participants received the site's standard practice treatment during the surgical procedure. Post-surgery, each participant was to undergo 78 weeks of follow-up for assessment of efficacy and safety.
- SRM003: Participants received a single application of 3 sponges at the time of the AVG placement: 1 sponge was wrapped around the venous anastomosis; another sponge was placed longitudinally on the vein segment, immediately distal to the venous anastomosis; and the remaining sponge was wrapped around the arterial anastomosis. Subjects were not permitted to undergo additional applications with SRM003 sponges after the initial application. After surgery, subjects were to undergo assessments during the 78-week follow-up period.
Period: Overall Study
Arm/Group | Participating Site's Standard Practice | SRM003
Started | 14 | 18
Completed | 0 | 0
Not Completed | 14 | 18
Not completed — Adverse Event | 2 | 1
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Study terminated by sponsor | 9 | 14
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other unspecified | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat population, defined as all randomly assigned participants regardless of the treatment received or having post-baseline outcome data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Participating Site's Standard Practice | SRM003 | Total
Number analyzed (Participants) | 14 | 18 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (10.0) | 60.9 (7.9) | 61.7 (8.8)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 9 | 12 | 21
  ≥65 years | 5 | 6 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Loss of Unassisted Primary Patency
Description: Unassisted primary patency (intervention--free access survival) was defined as the duration of time in days from the date of randomization (arteriovenous graft [AVG] placement) until the first date of (a) any intervention designed to establish, maintain, or restore patency, (b) occlusion (commonly due to thrombosis), or (c) access abandonment. Assessment of AVG patency was evaluated during physical examination of the subject's AVG at each visit and through ongoing AVG monitoring and surveillance according to each participating site's standard practice. It was recommended to follow the National Kidney Foundation Kidney guidelines (National Kidney Foundation 2006) on appropriate management and treatment of AVG complications to improve the function and longevity of the vascular access.
Time Frame: Up to 78 weeks after surgery
Population: The Intent to-Treat (ITT) population, defined as all randomly assigned participants regardless of the treatment received or having post-baseline outcome data.
Measure: Number; unit: percentage of participants
Arm/Group | Participating Site's Standard Practice | SRM003
Number analyzed (Participants) | 14 | 18
percentage of participants | 35.7 | 66.7
Statistical Analysis 1: Comparison: Participating Site's Standard Practice vs SRM003; Analysis of time to loss of patency; Test type: Superiority or Other; p = 0.138, Log Rank — p-value based on log rank test stratified by diabetic status at surgery comparing the 2 treatment groups

2. Secondary Outcome: Percentage of Participants With Loss of Assisted Primary Patency
Description: Assisted primary patency (thrombosis--free access survival) was defined as the duration of time in days from the date of randomization (AVG placement) until the first date of (a) occlusion (commonly due to thrombosis) or (b) access abandonment. Assessment of AVG patency was evaluated during physical examination of the subject's AVG at each visit and through ongoing AVG monitoring and surveillance according to each participating site's standard practice. It was recommended to follow the National Kidney Foundation Kidney guidelines (National Kidney Foundation 2006) on appropriate management and treatment of AVG complications to improve the function and longevity of the vascular access.
Time Frame: Up to 78 weeks after surgery
Population: The ITT population, defined as all randomly assigned participants regardless of the treatment received or having post-baseline outcome data.
Measure: Number; unit: percentage of participants
Arm/Group | Participating Site's Standard Practice | SRM003
Number analyzed (Participants) | 14 | 18
percentage of participants | 28.6 | 55.6
Statistical Analysis 1: Comparison: Participating Site's Standard Practice vs SRM003; Analysis of time to loss of patency; Test type: Superiority or Other; p = 0.312, Log Rank — p-value based on log-rank test stratified by diabetic status at surgery comparing the 2 treatment groups

3. Secondary Outcome: Percentage of Participants With Loss of Secondary Patency
Description: Secondary patency (access survival until abandonment) was defined as the duration of time in days from the date of randomization (AVG placement) until the date of access abandonment. Assessment of AVG patency was evaluated during physical examination of the subject's AVG at each visit and through ongoing AVG monitoring and surveillance according to each participating site's standard practice. It was recommended to follow the National Kidney Foundation Kidney guidelines (National Kidney Foundation 2006) on appropriate management and treatment of AVG complications to improve the function and longevity of the vascular access.
Time Frame: Up to 78 weeks after surgery
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Participating Site's Standard Practice | SRM003
Number analyzed (Participants) | 14 | 18
percentage of participants | 7.1 | 27.8
Statistical Analysis 1: Comparison: Participating Site's Standard Practice vs SRM003; Analysis of time to loss of patency; Test type: Superiority or Other; p = 0.093, Log Rank — p-value based on log-rank test stratified by diabetic status at surgery comparing the 2 treatment groups

4. Secondary Outcome: Number of Interventions to Establish, Maintain, or Restore Patency
Description: The total numbers of interventions to establish, maintain, or restore patency was assessed at the Week 26 visit.
Time Frame: 26 weeks after surgery
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: interventions
Arm/Group | Participating Site's Standard Practice | SRM003
Number analyzed (Participants) | 14 | 18
interventions | 0.7 (2.16) | 0.9 (1.00)
Statistical Analysis 1: Comparison: Participating Site's Standard Practice vs SRM003; Test type: Superiority or Other; Mean treatment difference = 0.230, 95% CI 2-sided [-0.942 to 1.402]

ADVERSE EVENTS:
Description: Treatment emergent adverse events are presented for the safety population, defined as all randomly assigned participants who received either SRM003 treatment or participating sites' standard practice treatments.
Arm/Group | Participating Site's Standard Practice | SRM003
Serious Adverse Events (participants affected / at risk) | 10/14 | 10/18
Other Adverse Events (participants affected / at risk) | 13/14 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participating Site's Standard Practice (N=14) | SRM003 (N=18)
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Arteriovenous graft site infection (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Arteriovenous graft site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Staphylococcus test positive (Investigations) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain compression (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Dry gangrene (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Steal syndrome (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Venous stenosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participating Site's Standard Practice (N=14) | SRM003 (N=18)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Local swelling (General disorders) | 0 (0) | 1 (1)
Medical device complication (General disorders) | 1 (1) | 2 (2)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Ulcer (General disorders) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Haemodialysis complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incision site hypoaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) | 3 (7)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 4 (5) | 5 (6)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Body temperature decreased (Investigations) | 1 (1) | 0 (0)
Brain natriuretic peptide increased (Investigations) | 1 (1) | 0 (0)
Grip strength decreased (Investigations) | 1 (1) | 0 (0)
Human chorionic gonadotropin positive (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Finger deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (3)
Cerebrovascular accident (Nervous system disorders) | 1 (2) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 4 (5) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ingrown hair (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arteriovenous graft (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Dialysis (Surgical and medical procedures) | 0 (0) | 1 (1)
Thrombectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 2 (3) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0)
Vasospasm (Vascular disorders) | 0 (0) | 1 (1)
Venous stenosis (Vascular disorders) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
Study was discontinued early due to Sponsor decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually